CLINICAL TRIAL: NCT04120727
Title: Evaluation of the Brakes and Levers on the Use of an E-health Therapeutic Education Application for Osteoarthritis Patients
Brief Title: Evaluation of the Brakes and Levers on the Use of an E-health Application for Osteoarthritis Patients
Acronym: ARTHe-1
Status: Completed | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: BPIfrance (Other); Innovatherm (Industry); La région Auvergne-Rhône-Alpes (Unknown); les thermes de Caleden (Unknown); Les thermes de Royat (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2019 ARTHe-1
Record Dates: First submitted 2019-10-08; First posted 2019-10-09 (Actual); Last update posted 2019-10-09 (Actual); Status verified 2019-07

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis; eHealth; therapeutic education; Connected objects
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patient: patients with predominant osteoarthritis of the knees
- Health professionals: health professionals with a link to osteoarthritis (physical and rehabilitation doctor, Rheumatologist, Physiotherapist, family doctor, pharmacist, Adapted physical activity teacher)

SUMMARY:
Osteoarthritis is the most common articular disease affecting the joint in a comprehensive and progressive manner. It is a chronic pathology correlated with age since nearly one in two adults is affected by osteoarthritis. The care of osteoarthritis is based on pharmacological and non-pharmacological treatment. The latest recommendations support the non-pharmacological part including regular physical activity, therapeutic education and weight loss. Today tools are lacking for the patient and the practitioner to ensure long-term motivation and support.

Connected objects, as future-oriented tools, are a customizable way to meet the expectations of both patients and professionals. The main objective of this study is to analyze the expectations regarding the use of a smartphone application for monitoring and support in the practice of exercises and regular physical activity in patients osteoarthritic.

The secondary objective is to collect information on the use of connected objects dedicated to the management of osteoarthritis by patients and health professionals.

DETAILED DESCRIPTION:
This study is aimed at patients with predominant knee osteoarthritis and health professionals with a link to the pathology.

A semi-directed interview according to a pre-established interview guide will be performed. Interviews are conducted by trained professionals and recorded with a dictaphone. Self-questionnaires are submitted to the patient after the interview.

The recordings are transcribed as quickly as possible in text format. The verbatim will then be coded (axial coding) then grouped by categories and then by themes.

The objective is to determine the expectations of patients and health professionals regarding a smartphone application dedicated to osteoarthritis.

This study will serve as a basis for designing a tool of this type to improve the long-term management of osteoarthritis.

ELIGIBILITY:
Inclusion Criteria for Patient :

* Patient with osteoarthritis according to the criteria of the ACR (American College of Rheumatology), symptomatic and diagnosed in advance of inclusion by a specialist physician or not

Inclusion Criteria for Professional :

-Selected health professionals must be in practice at the time of inclusion. General practitioners, MPR (Physical and Rehabilitation Medicine), rheumatologists, physiotherapists, APA (Professor of Adapted Physical Activity) and pharmacists caring for arthrosic patients, either salaried or liberal and on the volunteering base.

Exclusion Criteria:

* Patients who do not meet the diagnostic criteria of the ACR (American College of Rheumatology)
* Patients with comprehension disorders which make it impossible to maintain and fill out questionnaires.
* Refusal to participate or already included in a therapeutic education workshop.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients : Adult with osteoarthritis Healt professionnal : Health professionals in contact with arthrostic patients
Sampling Method: Non-Probability Sample
Enrollment: 32 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Brakes and levers on the use of an e-health therapeutic education tool for arthrosic patients | Day 1
  A qualitative study that aims to target expectations of an e-health therapeutic education application. An interview (individual semi-directed interview method) is scheduled to be conducted with patients and practitioners lasting 20 to 40 minutes. This interview is divided into 3 items: daily physical activity, opinion on connected objects dedicated to health, key points that should be included in the application

SECONDARY OUTCOMES:
socio-demographic questionnaire | Day 1
  This questionnaire will help to categorized subjects in sub-group
Measure of Kinesiophobia | Day 1
  TSK (Tampa Scale of Kinesiophobia) scale will be used
Measure of Knee injury | Day 1
  KOOS (Knee injury and Osteoarthritis Outcome Score) scale will be used
Measure of physical activity perception | Day 1
  EPAP (Evaluation of perception of physical activity) scale will be used

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Thermes CALEDEN - Société thermale de Chaudes Aigues, Chaudes-Aigues, Auvergne-Rhône-Alpes
  - CHU Gabriel Montpied, Clermont-Ferrand, Auvergne-Rhône-Alpes
  - Thermes de ROYAT - Régie Municipale des eaux minérales de Royat / SPIC, Royat, Auvergne-Rhône-Alpes